CLINICAL TRIAL: NCT02799771
Title: Observational Study of Incident Patients With Pre Capillary Pulmonary Hypertension and Interstitial Lung Disease
Brief Title: HYPID (Pulmonary Hypertension in Interstitial Lung Disease) EXTENSION
Acronym: HYPID-2
Status: Completed | Type: Observational
Sponsor: Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Vincent COTTIN, Professor Vincent COTTIN, Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires
Other Study IDs: GERMOP- 005
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Arterial Hypertension; Diffuse Interstitial Lung Disease
Keywords: Pulmonary arterial hypertension; Interstitial lung disease at HRCT
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
HYPID-2 study is an extension of HYPID study (NCT01443598) :

HYPID-2 is also an observational and prospective study of patients with interstitial lung disease and pre capillary hypertension diagnosed by right heart sided catheterization.

It concerns only incident patients (i.e patients included within 6 months after PH diagnosis) whereas HYPID concerned prevalent and incident cases.

The primary aim is the same than HYPID : identify prognostic factors

DETAILED DESCRIPTION:
Pre capillary pulmonary hypertension (PH) may be present in patients with diffuse interstitial lung disease.

In this context, PH represents an important factor of morbidity and mortality for these patients.

As in HYPID, the main purpose of HYPID-2 is to determine predictive factors of mortality within this cohort of incident patients (i.e patients included within 6 months after PH diagnosis).

In order to reach that aim,the study includes an evaluation based on exams conducted for the routine follow-up of incident patients.

Each incident patient will be followed during 2 years at least.

ELIGIBILITY:
Inclusion Criteria:

Patients newly diagnosed with:

* Pre capillary pulmonary hypertension at right heart sided catheterization with: mPAP > or = 25 mmHg, PCWP < or = 15 mmHg
* Interstitial lung disease with diffuse infiltrative opacities on chest CT scan

Exclusion Criteria:

* Pulmonary hypertension related to a thromboembolic disease
* Respiratory disease other than diffuse interstitial lung disease
* Any etiological factor of pulmonary arterial hypertension based on NICE 2013 classification other than diffuse interstitial lung disease
* Any progressive disease associated to a life expectancy less than 6 months other than pulmonary hypertension, diffuse interstitial lung disease and respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident patients with pre capillary pulmonary hypertension and interstitial lung disease at HRCT
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Determine predictive factors of mortality

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Time to death or 10% decline in FVC
Response to therapy | 2 years
  Proposition of patients with 10% or more decline in PVR

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COTTIN, MD, Principal Investigator — Hospices civils de Lyon / Université Lyon I
Locations (1):
- Louis Pradel Hospital (Bâtiment A4), Lyon, Bron, France

REFERENCES:
- See also: website National French Reference Center for rare lung diseases — http://maladies-pulmonaires-rares.fr/